CLINICAL TRIAL: NCT02976506
Title: Safety of an Unsupervised Physical Activity Program and Effects Over Blood Pressure, Physical Fitness and Quality of Life of Elderly Hypertensive Patients
Brief Title: Unsupervised Physical Activity in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Patricia Silva Carneiro, Principal Investigator, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30847614.6.0000.5078
Record Dates: First submitted 2016-11-14; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Elderly; Hypertension; Physical Conditioning
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Physical Fitness; Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unsupervised exercise program (Experimental): To verify the interference of an unsupervised exercise program on blood pressure, physical fitness, quality of life and safety in elderly hypertensive patients. Participants were divided into the study group or control group
  Interventions: Behavioral: Unsupervised exercise program
- Physical fitness and quality of life (Experimental): To verify the interference of a walking program on physical fitness and quality of life.
  Interventions: Behavioral: Physical fitness and quality of life

INTERVENTIONS:
Behavioral: Unsupervised exercise program — Both control and intervention group undergo clinical evaluation, and anthropometric measurements, blood pressure (casual and ambulatory blood pressure monitoring), physical and laboratorial tests, and the assesment of Quality of Life by Questionnaire SF-36 were done at the beginning and the end of the study.After a period of 12 weeks of unsupervised walking program in which participants were asked to do it three times a week at least, at a moderate intensity (40 to < 60% of heart rate reserve), all participants underwent a complete re-evaluation to compare the results obtained with the proposed program. Data were analyzed using SPPS, v.23.0.
  Other Names: interference on blood pressure
  Arms: Unsupervised exercise program
Behavioral: Physical fitness and quality of life — Both control and intervention group undergo clinical evaluation, and anthropometric measurements, blood pressure (casual and ambulatory blood pressure monitoring), physical and laboratorial tests, and the assesment of Quality of Life by Questionnaire SF-36 were done at the beginning and the end of the study.After a period of 12 weeks of unsupervised walking program in which participants were asked to do it three times a week at least, at a moderate intensity (40 to < 60% of heart rate reserve), all participants underwent a complete re-evaluation to compare the results obtained with the proposed program. Data were analyzed using SPPS, v.23.0.
  Arms: Physical fitness and quality of life

SUMMARY:
To evaluate safety and the effects of a unsupervised physical activity program (USPAP) over blood pressure (BP), physical fitness (PF) and quality of life (QL) of elderly hypertensive patients.

DETAILED DESCRIPTION:
The present study was approved by the Human and Animal Ethics Committee of the institution and the participants were only randomized to participate after having signed the informed consent form.

A population of elderly hypertensive patients registered at a reference center for hypertension treatment was selected. The sample size was calculated considering a test power of 80% with significance level of 5% and estimating a difference to be observed within the BP values of 7 mmHg for systolic blood pressure (SBP) and 4 mmHg for diastolic blood pressure (DBP). The sample calculated was 25 participants in each group being selected 20% more in case of losses.

An electronic chart was created with numbers for the patients that were randomized into control (CG) and intervention groups (IG).

The IG was included in an USPAP and the control group was kept under the usual care of the service that includes orientation to perform PA according to the World Health Organization recommendations.

Before the beginning of the protocol clinical and laboratorial data collected included: weight, height, waist circumference, fasting glucose, hemoglobin A1C and lipid profile.

In addition to that health-related quality of life was assessed with the Short Form 36-item Health Survey (SF-36). The SF-36 Questionnaire includes one multi-item scale that assesses eight health concepts: 1) functional capacity; 2) physical aspects; 3) pain; 4) general health status; 5) vitality; 6) social aspects; 7) emotional aspects; and 8) mental health. The score of each health concept ranges from 0 to 100, in which zero means the worst general health state and one hundred the best health state.

All patients underwent physical tests to evaluate their physical fitness: cardiorespiratory fitness test (Cooper Test) and abdominal resistance test. Patients were classified according to the Physical Aptitude Classification Tables for Users of Public Parks.

The BP was assessed with office BP measurements using OMRON - HEM 705 CP® semi-automatic devices according to the VI Brazilian Hypertension Guidelines (BHG). Home blood pressure was also performed following the same technics of office measurements and according to the III Brazilian Guidelines of Home Blood Pressure Monitoring with 3 measurements in the morning fasting and 3 at night before dinner in four consecutive days.

The physical activity prescriptions were individualized so that the patients would have no doubts regarding execution when performing the exercise without the presence of the prescribing professional. The prescribed physical activity was aerobic and walking was the chosen one. The activity was prescribed in a planned, structured and repetitive way aiming to maintain or improve one or more components of physical fitness. To achieve those goals patients attended to 2 supervised sessions that took place in a one week period in non-consecutive days. They were instructed to perform training at least 3 times a week during 30 minutes or more with a moderate intensity of 40 to 60% of their reserve heart rate which mean walking slightly breathless but being able to pronounce complete phrases according to the VI BHG recommendations. The total number of sessions prescribed was 36 throughout the 12 weeks. The minimum of 30 sessions was needed so the results could be validated.

Health educational strategies were used simultaneously to data collection to improve adherence of both groups. Motivational actions were used specific for the IG. Weekly phone calls were carried out to the IG in order to know about the number of sessions performed that week, the duration of the practice and the total number of steps of each session. All participants received a pedometer and a diary to register activities.

Safety was assessed considering: need to interrupt training due to lesions, falls, incapacitating pain or acute events related to training that would require medical assistance.

After 12 weeks all participants were reevaluated and all procedures were repeated to evaluate the effects of the intervention.

Data collected was analyzed with software Statistical Package of Social Science, version 23.0, Chicago, USA. Qualitative variables were presented in absolute numbers and percentages with the comparison between them being made with Qui Square Test or Exact Fisher Test. Proportion comparison in the groups was performed applying Wilcoxon Test. Quantitative variables were initially analyzed in terms of its distribution with Shapiro-Wilk test. Mean variables comparison was performed with T-Student test for paired and unpaired samples. The results were presented as mean values and standard deviation and p value < 0,05 was considered significant.

ELIGIBILITY:
The inclusion criteria were:

* 60 years old or more, stable BP on the last three months, no changes on pharmacological treatment over the last six months and a sedentary behavior (non-participation in any kind of physical activity for at least 2 months).

The exclusion criteria considered were:

* uncontrolled diabetes
* congestive heart failure
* acute myocardial infarction in the last six months
* stroke in the last six months or under rehabilitation
* previously diagnosed chronic renal failure
* acute infectious diseases
* recent systemic or pulmonary embolism
* pulmonary hypertension
* BP higher than 159 x 99 mmHg
* neuromuscular
* musculoskeletal or articular disorders diagnosed and not treated
* clinical evaluation restraining PA
* any situation preventing the patient from walk. Those criteria were verified in patients' medical charts.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lower Blood Pressure and or keeping it under control | 12 weeks

SECONDARY OUTCOMES:
Improve Cardiorespiratory fitness. | 12 weeks
  Cooper Test (before and after the intervention).
Improve abdominal strength. | 12 weeks
  Abdominal resistance test before and after the intervention.
Quality of life | 12 weeks
  SF-36 questionnaire before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension League, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
OPEN ACCESS